CLINICAL TRIAL: NCT01909882
Title: The Effect of Family Members' Massage Therapy on Vital Signs and Glasgow Coma Scale Score of Patients Hospitalized in Intensive Care Unit: A Triple-blinded Randomized Controlled Clinical Trial Study
Brief Title: Effect of Family Member's Massage Therapy on the Vital Signs and Glasgow Coma Scale Score
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baqiyatallah Medical Sciences University (Other)
Collaborators: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Amir Vahedian-Azimi, Dr, Baqiyatallah Medical Sciences University
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Supportive Care
Other Study IDs: Massage therapy
Record Dates: First submitted 2013-07-22; First posted 2013-07-29 (Estimated); Last update posted 2013-07-29 (Estimated); Status verified 2012-08

CONDITIONS: Trauma
Keywords: Family member's massage therapy; Vital signs; Glasgow coma scale; Intensive care unit; Randomized controlled Clinical Trial; Iran
MeSH Terms: conditions — Wounds and Injuries | interventions — Massage

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Family member's massage therapy (Other): Family member's massage therapy
  Interventions: Other: Massage therapy

INTERVENTIONS:
Other: Massage therapy — One session of massage therapy (for 60 minutes) was done by the patient's family member. Almond oil was used for effleurage and massage facilitation. Back, shoulder deltoid muscles, front and posterior parts of legs, arms, forearms, front and back parts of thighs, palms and fingers, metatarsus, front and back of feet and toes, belly and chest, auxiliaries and neck muscles of the patients were massaged. Massage techniques used included static massage, surface tension techniques, stretching massage, superficial lymph unload, transverse friction techniques, and myofacial releasing techniques. All the massage sessions were conducted in the morning shifts. For the control group, there was no intervention and patients just received the routine care of the unit.

SUMMARY:
The effect of family member's massage therapy on the Vital signs and Glasgow Coma Scale Score of hospitalized patients in Intensive Care Unit: A Triple-blinded Randomized controlled Clinical Trial Study

DETAILED DESCRIPTION:
Aims and objectives: To determine the effects of family member's massage therapy on the Vital signs and Glasgow Coma Scale Score of hospitalized patients in Intensive Care Unit.

Background: Unalleviated complications related to hospitalization including stress, anxiety, pain, and fear can easily impacts on different systems including brain and stimulates sympatric nerves and as a result causes instabilities in vital signs and deterioration in consciousness level. Alternative and complementary therapies including therapeutic massage have been used to decrease the mentioned side effects.

Design: A Triple-blinded Randomized controlled Clinical Trial Methods: All prolonged hospitalized patients and their families (45 patients and 45 family members in each group) were selected consecutively among the patients admitted in ICU. Data collection tool consisted of two parts. The first part included demographic data (age, mar¬ital status and Body Max Index) and the second part included a checklist to record the patient's vital signs (systolic blood pressure, diastolic blood pressure, respiratory rate, and pulse rate). All measurements were conducted in same time in both groups as follow: before the intervention (the whole massage therapy), one hour, two hours, three hours, and four hours. Collected data was analyzed using descriptive and analytical statistics utilizing SPSS 11.5 software.

Keywords: Family member's massage therapy; Vital signs; Glasgow coma scale; Intensive care unit; Randomized controlled Clinical Trial; Iran.

ELIGIBILITY:
Inclusion Criteria:

* more than 10-day hospitalization, hemodynamic stability, having the Glasgow coma scale score between 7 to 12, intra cranial pressure less than 20 mmHg, no limitation or contraindication for changing in body position (including active bleeding or flail chest) and body massage (such as advanced burn degrees, severe dyspnea, fever, etc) and willing to participate in the study

Exclusion Criteria:

* Any factors which violate inclusion criteria

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Systolic Blood Pressure | 1 year
  Change in Systolic Blood Pressure

SECONDARY OUTCOMES:
Diastolic Blood Pressure | 1 year
  change in diastolic blood pressure
Respiratory Rate | 1 year
  change in respiratory rate
Pulse Rate | 1 year
  change in pulse rate
Glasgow Coma Scale | 1 year
  change in Glasgow Coma Scale

CONTACTS AND LOCATIONS:
Overall Officials: amir vahedian-azimi, professor, Principal Investigator — BMSU
Locations (1):
- Shariati hospital, Tehran, Tehran Province, Iran